CLINICAL TRIAL: NCT01734616
Title: Dysfunction of Nutritive Blood Flow as a Determinant of Anabolic Resistance in Older People
Acronym: Dunhill01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: F/3/2009
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Regional Blood Flow
Keywords: Microvascular; Muscle; Nutrition; Exercise; Ageing
MeSH Terms: conditions — Motor Activity | interventions — Chocolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Young (No Intervention): Young subjects to be controlled to older individuals with interventions
- Old (No Intervention): Older individuals to compare to young and other older intervention groups
- Old Exercise (Experimental): Older individuals studied after an intervention of 20 weeks fully-supervised resistance exercise training
  Interventions: Behavioral: Old Exercise
- Old Acute Cocoa (Experimental): Older individuals studied with the addition of cocoa flavanols during their acute study
  Interventions: Dietary Supplement: Old Acute Cocoa
- Old 7 Day Cocoa (Experimental): Older individuals studied after 7 day supplementation of cocoa flavanols
  Interventions: Dietary Supplement: Old 7 Day Cocoa

INTERVENTIONS:
Behavioral: Old Exercise
  Arms: Old Exercise
Dietary Supplement: Old Acute Cocoa
  Arms: Old Acute Cocoa
Dietary Supplement: Old 7 Day Cocoa
  Arms: Old 7 Day Cocoa

SUMMARY:
With age, muscles tend to waste at 0.5-1% per year, so that an 80 year old may have only 70% of the muscle possessed at 50. Muscle loss makes it harder to carry out tasks that require strength, keep the body balanced and continue activity for a prolonged period, which together may contribute to a loss of independence and an increased risk of falls. The cause of some of this muscle loss with ageing appears to be a reduction in muscle building in response to food. The known decreased limb blood flow in ageing muscle may go some way to explain this as there may be less nutrient delivery to the muscles. The investigators want to test if the known decrease in limb blood flow with age is matched with a decrease in the proportion of blood being delivered directly to the muscles, rather than fat and connective tissue. If so the investigators expect to see an improvement in the ability of muscles to maintain themselves via better capture of amino acids into protein. The investigators also want to test if 20 weeks resistance exercise training or drinking a cocktail of mixture of high flavanol cocoa (which can increase blood flow) and vitamin C can improve limb blood flow to older muscles and help reduce muscle wasting.

DETAILED DESCRIPTION:
By 2020, 20% of the UK population will be over 65 y. Muscle mass is a strong predictor of healthy ageing and longevity. Basal limb blood flow decreases with advancing age; reduced limb perfusion may contribute to sarcopenia, the undesirable loss of muscle mass that accompanies advancing age. The investigators previous work has shown that there are deficits in the mechanisms of muscle protein synthesis in older people, but why these exist and how they may be countered is still unknown. After normal feeding, increased amino acid availability (stimulating muscle protein synthesis) and insulin availability (inhibiting muscle protein breakdown) do have good effects in the muscle of older people but not to the same extent as in the young; the investigators call this "anabolic resistance". The investigators have recently shown that leg blood flow in elderly people is lower than in the young at rest in the basal state and also at rest up to 2.5 hours after food and or food + exercise. The matching of blood flow and metabolism is advantageous for skeletal muscle, in marrying demands for oxygen and nutrients to their delivery; the reduced limb perfusion in the older people may contribute to an inability to maintain muscle mass with ageing. The investigators have recently shown that resistance training markedly improves leg blood flow responses in elderly persons. They believe a major benefit of resistance exercise is to increase endothelium dependent vasodilation in response to feeding and moderate exercise, but this needs to be proved. It is becoming recognised that it is not only "bulk" limb blood flow that may be important in muscle nutrient uptake but that so called 'nutritive' blood flow is an important determinant. Recent work suggests that bulk limb flow is not only partitioned between skin, bone and muscle but even within muscle is partitioned between 'nutritive' and 'non-nutritive'. The nutritive route has intimate contact with muscle cells while the non-nutritive route acts as a vascular shunt and is thought to be, at least in part, via vessels that nourish fat and connective tissue cells. Nutritive flow may be the component of flow which is most susceptible to dysfunction5 (e.g. with type 2 diabetes and obesity) but may also be the most susceptible to improvement by accustomed exercise and possibly nutraceutical treatment.

The investigators will test the hypotheses: (1) muscle nutritive blood flow is a determinant of protein balance, with pharmacologically induced vasodilation acutely stimulating muscle synthesis and reducing breakdown, (2) low nutritive flow in elderly people contributes to anabolic resistance and can be ameliorated by resistance training or nutraceutical flow enhancers.

The investigators wish to study 50 healthy volunteer subjects (not NHS patients) as follows: 18-28 y men (10) and 65-75 y men (40) of comparable body mass index (24-28 kg•m2) all of whom are sedentary and normally undertake no customary resistance training. The investigators have data suggesting sexual dimorphism of anabolic responses to feeding in older subjects so will restrict studies to men only. After obtaining written consent, all subjects will undergo a medical examination, activity questionnaire and DEXA scan. Ten elderly men will undergo a single acute study. In addition the investigators will study 10 young men under the same conditions. Ten more elderly men will undergo an acute study after 20 weeks of supervised whole-body resistance training, as is current practice at a gym site in Derby. Ten more elderly men will undergo a single acute study in which they are given, in addition to the standard acute study protocol 3 drinks of high flavanol cocoa and 3 x 500 mg of vitamin C. If a positive acute effect of the drinks is observed the final ten elderly men will undergo an acute study after a week of ingesting 3 high flavanol cocoa + 1000 mg of vitamin C per day. To optimise details of study conditions the investigators will also study up to 10 normal healthy volunteers 18-75 y simply with the CEUS contrast agent and methacholine infusions, without any blood sampling or biopsies.

Subjects fasted overnight will receive primed constant intravenous (antecubital vein) infusions of stable isotope labelled amino acids for the duration of the study and blood samples will be taken from an arterial cannula and two femoral venous cannulae at regular intervals to quantify tracer enrichment and measure glucose uptake and insulin. In the first phase of the study, subjects' bulk femoral artery blood flow will be measured at 50, 70, 90 and 110 min by Doppler Ultrasound (USS). Nutritive blood flow will be measured in a defined area of the quadriceps in the control leg by Contrast Enhanced Ultrasound (CEUS) using the Phillips iU22 at 110 min. This involves a single intravenous administration of SonoVue® contrast agent. At 120 min the second phase of the study will begin with a dextrose and mixed amino acid intravenous infusion (antecubital vein) for the remainder of the study. Methacholine chloride (Provocholine®; Methapharm Inc.) in NaCl (0.9%, prepared by QMC pharmacy)will be infused (at 2-12 µg/min) into one femoral artery to double femoral artery flow at 150 min. Bulk femoral artery flow will again be measured (Doppler Ultrasound), this time in both legs at 170, 190, 210 and 230 min. Nutritive flow will be measured for a second time, in both legs by CEUS at 230 min. Four muscle biopsies (150-300 mg) of vastus lateralis will be taken according to the protocol and snap-frozen in liquid nitrogen.

The end points will be i. muscle protein synthesis, ii. muscle protein breakdown, iii. bulk femoral blood flow and iv. nutritive femoral blood flow in subjects of different ages or following different exercise or nutraceutical intervention. A power calculation suggests that this study will need 10 subjects per group to detect (with α of 0.05 and β of 0.85) a 25 % difference between groups in biological variables, results the investigators have been able to achieve for similar work in the past.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers aged 18-28 or 65-75

Exclusion Criteria:

* Overt muscle wasting i.e. muscle mass is more than 1 standard deviation below normal muscle or FFM for age
* A BMI < 24 or > 28 kg•m2.
* Active cardiovascular disease: uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt or recent cardiac event
* Individuals taking beta-adrenergic blocking agents.
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial).
* Respiratory disease including pulmonary hypertension, COPD, asthma or an FEV1 less than 1.5 l.
* Metabolic disease: hyper and hypo parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes.
* Active inflammatory bowel disease, or renal disease,
* Malignancy
* Recent steroid treatment (within 6 mo), or hormone replacement therapy.
* Clotting dysfunction
* Musculoskeletal or neurological disorders.
* Family history of early (<55y) death from cardiovascular disease
* Known sensitivity to Definity or methacholine

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Microvascular blood volume in response to feeding | September 2009 - August 2012
  The final study participant was completed and all microvascular blood volume data analysed by August 2012. This outcome measure is applicable to all arms of this study and refers to responsiveness to a 2 hour feed protocol.

SECONDARY OUTCOMES:
Muscle protein metabolism in response to feeding | January - October 2012
  Muscle protein metabolism (synthesis and breakdown) in response to feeding in young and older individuals and in older individuals after exercise or nutraceutical intervention. This outcome measure could only be assessed after all studies were completed to ensure standardization of mass-spectrometry measurements between the groups.

OTHER OUTCOMES:
Molecular pathways regulating muscle microvascular blood volume | August 2012 - August 2013
  This outcome measure was not able to be analysed prior to completion of all studied and the subsequent primary and secondary outcome measures as molecular targets of interest were dependent upon these results. This analysis has began and should be complete by August 2013.

CONTACTS AND LOCATIONS:
Overall Officials: John P Williams, PhD, MD, Principal Investigator — University of Nottingham; Bethan E Phillips, PhD, Study Director — University of Nottingham
Locations (1):
- Clinical Physiology Laboratory, Graduate Entry Medical School, University of Nottingham, Royal Derby Hospital, Derby, Derbyshire, United Kingdom

REFERENCES:
- [Background] Phillips B, Williams J, Atherton P, Smith K, Hildebrandt W, Rankin D, Greenhaff P, Macdonald I, Rennie MJ. Resistance exercise training improves age-related declines in leg vascular conductance and rejuvenates acute leg blood flow responses to feeding and exercise. J Appl Physiol (1985). 2012 Feb;112(3):347-53. doi: 10.1152/japplphysiol.01031.2011. Epub 2011 Oct 13. PMID 21998269